CLINICAL TRIAL: NCT04338126
Title: Exploratory Studies of the Effect of Tranexamic Acid Treatment on the Progression of COVID19 in Inpatients
Brief Title: Tranexamic Acid (TXA) and Corona Virus 2019 (COVID19) in Inpatients
Acronym: TCInpatient
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to ongoing vaccination efforts, feasibility for recruitment is low
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Timothy Ness, MD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TXACOVID2
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19 | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double blind comparison
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacy prepares medications that are coded
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid Treatment (Experimental): Oral dosing of tranexamic acid at dose of 1300 mg p.o. three times per day x 5 days; alternative dosing intravenously with loading dose of 10 mg/kg followed by 1 mg/kg/hr infusion x 5 days
  Interventions: Drug: Tranexamic acid
- Placebo Treatment (Placebo Comparator): 2 tablets of placebo three times per day x 5 days; alternative dosing intravenous normal saline at volumes similar to those use for experimental arm
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Tranexamic acid — previously described
  Arms: Tranexamic Acid Treatment
Drug: Placebo oral tablet — previously described
  Arms: Placebo Treatment

SUMMARY:
A controlled trial of the drug tranexamic acid (TXA) in inpatients recently admitted to the hospital with the diagnosis of COVID19. It is hypothesized that TXA will reduce the infectivity and virulence of the virus.

DETAILED DESCRIPTION:
A recent report in Physiological Reviews proposed that the endogenous protease plasmin acts on COVID19 virus by cleaving a newly inserted furin site in the S protein portion of the virus resulting in increased infectivity and virulence. Patients with hypertension, diabetes, coronary artery disease, cerebrovascular illness, lung disease and kidney dysfunction commonly have elevated levels of plasmin/plasminogen and it was proposed that this may be the mechanism for poorer outcomes in patients with these co-morbidities. A logical treatment that might blunt this process would be the inhibition of the conversion of plasminogen to plasmin. Fortunately, there is an inexpensive, commonly used drug, tranexamic acid (TXA) which suppresses this conversion and could be re-purposed for the treatment of COVID19. TXA is a synthetic analog of the amino acid lysine which reversibly binds four to five lysine receptor sites on plasminogen. This reduces conversion of plasminogen to plasmin, and is normally used to prevent fibrin degradation. TXA is FDA approved for treatment of heavy menstrual bleeding (typical dose 1300 mg p.o. three times per day x 5 days) and off-label use for many other indications. TXA is used perioperatively as a standard-of-care at the University of Alabama at Birmingham (UAB) for orthopedic and cardiac bypass surgeries. At UAB, it is commonly employed in hemorrhaging trauma patients and currently is being studied for perioperative use in Cesarean section surgeries. It has also been utilized for spinal surgery, neurosurgery, orthognathic surgeries and even long term for the treatment of cosmetic dermatological disorders with a long track record of safety.

Given the potential benefit and limited toxicity of TXA it would appear warranted to perform a rapid randomized, double-blind placebo controlled exploratory trial at UAB in the treatment of the early phases of COVID19 to determine whether it reduces infectivity and virulence of the COVID19 virus as hypothesized. Involvement of each patient is only for 7 days before primary endpoints.

An exploratory, randomized, placebo-controlled, double-blind Phase 2 clinical trial in which study patients have just been admitted to the regular hospital (non-Intensive Care Unit; ICU) for the diagnosis of COVID19 is proposed. The overall goal of this exploratory study is to assess both safety and efficacy of 5 days of TXA versus placebo in the COVID19 population. All patients would also receive daily anticoagulation as directed by their primary care team. The primary endpoint for the study would be a need for transfer to an ICU. Contact would be daily and via remote processes. Care for the COVID19 patient would otherwise be standard of care and directed by the primary caretakers of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Positive COVID19 test
* Admission to hospital without immediate plans for Intensive Care Unit transfer
* Age >/= 19 y.o.

Exclusion Criteria:

* Allergic reaction to tranexamic acid
* History or active evidence of hypercoagulation disorders including but not limited to deep vein thrombosis, pulmonary hypertension, diffuse intravascular coagulopathy
* Preadmission anticoagulation
* History of GI bleeding
* History of seizures
* Cardiac or other vascular stents
* History of severe renal disease
* History of intracranial hemorrhage

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Admission to Intensive Care Unit | Randomization to 7 days after randomization
  Transfer to Intensive Care Unit for deteriorating clinical condition

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Ness, MD PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No